CLINICAL TRIAL: NCT06832345
Title: The Effect of Web-Based Training and Counseling Given to Caregivers on the Pressure Injury Risk, Level of Dependence-Independence, and Caregivers' Burden of Care in Bedridden Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Şerife Kelle Dikbaş, Phd Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: interventation
Record Dates: First submitted 2024-06-28; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Pressure Injury Prevention
Keywords: pressure injury prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventions to be applied to the experimental group (web-based training and consultancy ) (Other): Web-based education and counseling services will be provided as an intervention. Web-based education will be provided to the caregiver in the patient's room in two face-to-face sessions within forty-eight hours before the patient is discharged. Counseling will include telephone follow-up and home visits after discharge. Telephone follow-up will be done once a week, for a total of 8 times, and home visits will be done 3 times over an 8-week period. The results will be assessed using the Braden Pressure Injury Risk Scale, Barthell Index, and data collection tools for patients in the experimental group, and the Zarit Caregiver Burden Scale will be used for caregivers.
  Interventions: Other: Experimental group
- interventions to be applied to the control group (Other): Caregivers in the control group will receive routine nursing care and no intervention will be made. At the end of the study, the website and educational content will be shared with patients and their relatives.
  Interventions: Other: Experimental group

INTERVENTIONS:
Other: Experimental group — Web-based training will be shared with patient relatives before the patient is discharged. A home visit will be made 2-3 days after the patient is discharged. Data collection forms will be collected by the researcher at each home visit. A total of four home visits and eight telephone follow-ups will be made within two months.

SUMMARY:
Education and counseling of patients and caregivers, either face-to-face or using various communication technologies, are reported to have significant effects. Nurses are in a key position in the education and counseling of patients and their relatives for the prevention of pressure injury. Although the share of health technologies in the management of pressure injury is important, it is also important for nurses to use these technologies. Web-based education, which is a part of health technologies, is defined as an education and training program created by using the features of internet and computer technologies.

DETAILED DESCRIPTION:
To prevent pressure injuries; It has been determined that there are a limited number of studies in which training, telephone monitoring and counseling are provided to caregivers The originality of this study, which was conducted to evaluate the effect of web-based training given to caregivers on the pressure injury development of bedridden patients, addiction independence level and care burden of caregivers; The training is designed as web-based and creates a guide that caregivers can use during the care process.

ELIGIBILITY:
Inclusion Criteria:

The patient;

* Being over 18 years of age
* Being open to communication (Mini Mental Test Score >25 points),
* Medium or high risk according to the Braden pressure injury assessment scale (score ≤14 according to the Braden pressure injury risk assessment scale)
* Being at least a moderately dependent patient according to the Barthel Index (score ≤90 according to the Barthel Index) The caregiver;
* Being primarily responsible for patient care,
* Being over 18 years of age
* Having a family bond with the patient,
* No monthly fee for providing care, (except for those receiving a monthly care pension from the state)
* Lack of healthcare workers (physician, midwife, nurse),
* Ability to read and write,
* Having a smartphone and internet access,
* Accepting a home visit,
* There is no physical or psychiatric obstacle that prevents communication,

Exclusion Criteria:

The patient;

* Having cancer,
* Having an active skin disease,
* Blood glucose and blood pressure are not under control,
* Use of medication that may be associated with pressure injury (corticosteroid, immunosuppressive, sedative medication, antineoplastic medication, norepinephrine) is an exclusion criterion from the study.

Criteria for Exclusion from the Study The patient;

* The patient is hospitalized,
* The patient's exitus is a criterion for exclusion from the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Findings regarding sociodemographic characteristics | 8 weeks, "up to two months".
  Evaluation of data that may be related to pressure injuries for patients and caregivers.
  Data such as patient's age, height, weight, chronic diseases and data such as caregivers' age, inclination, and caregiving duration will be evaluated as averages and percentages.
Evaluation of the results regarding the patient's level of dependency and independence | 8 weeks, "up to two months".
  According to the total scores of the Barthell Life Activities Index; 0-20 points: "Fully dependent", 21-61 points: "Extremely dependent", 62-90 points: "Moderately dependent", 91-99 points: "Mildly dependent" and 100 points: "Fully independent"
Assessment of patient's pressure injury risk score | 8 weeks, "up to two months".
  According to the braden pressure injury risk assessment scale: The total scale score is between 6 and 23. As the scores from the scale decrease, the risk of developing a pressure injury increases. Individuals with a scale score of 12 and below are considered to be at high risk for developing a pressure injury, those with a score of 13-14 are considered to be at medium risk, and those with a score of 15-16 are considered to be at low risk. According to the inclusion criteria for this study, patients must be assessed as high and medium risk according to the Braden pressure injury risk assessment scale.
Results regarding the caregiver's care burden | 8 weeks, "up to two months".
  According to the zarit caregiver burden scale: If the resulting score is between 22-46 points, it is defined as 'light load', if it is between 47-55 points, it is defined as 'moderate load', and if it is between 56-110 points, it is defined as 'severe load'.

IPD SHARING:
Plan to Share IPD: No